CLINICAL TRIAL: NCT02647333
Title: Intervention With Omega Fatty Acids in High-risk Patients With Hypertriglyceridemic Waist
Brief Title: Intervention With Omega Fatty Acids in High-risk Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014/2336
Record Dates: First submitted 2015-09-09; First posted 2016-01-06 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids; Fish Oils; Fatty Acids, Omega-6

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 fatty acid (Experimental): Omega-3 fatty acids for 8 weeks, dosage are 3 and 4 g/day for women and men, respectively.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid
- Omega-6 fatty acid (Experimental): Omega-6 fatty acids for 8 weeks, dosage are 20 and 27 g/day for women and men, respectively.
  Interventions: Dietary Supplement: Omega-6 Fatty Acid

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — Experimental: Omega-3 fatty acid In the intervention period the participants will receive a daily supplement of omega-3 fatty acids for 8 weeks, where the dosage are 3 and 4 g/day for women and men, respectively. The omega-3 supplement is a hydrolyzed and reesterified TAG fish oil, containing 33 area percent eicosapentaenoic acid and 22 area percent docosahexaenoic acid.
  Other Names: Omega-3; N-3 Fatty Acid; Fish oil; N-3 PUFA
  Arms: Omega-3 fatty acid
Dietary Supplement: Omega-6 Fatty Acid — Experimental: Omega-6 fatty acid In the intervention period the participants will receive a daily supplement of omega-6 fatty acid for 8 weeks, where the dosage are 20 and 27 g/day for women and men, respectively. The omega-6 supplement is a high-quality organic, cold pressed and filtered safflower oil, containing 68-83% linoleic acid, 5-15% saturated fatty acid, 8-21% oleic acid, 0,0-0,5% ALA and maximum 2% other fatty acids.
  Other Names: Omega-6; N-6 Fatty Acid; N-6 PUFA
  Arms: Omega-6 fatty acid

SUMMARY:
In order to reduce cardiovascular risk, current European guidelines recommend a diet low on saturated fatty acid through replacement with polyunsaturated fatty acids (PUFA). Polyunsaturated fatty acids can be classified into omega-3 and omega-6. However the results from recent meta-analyses investigating coronary risk outcomes did not clearly support a low intake of saturated fatty acids and a high intake of omega-3 or omega-6. The aim of this study is to investigate the short term effects of a high intake of PUFAs on microvascular function, lipids, inflammation and other cardiovascular risk factors in inactive patients with increased waistline.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥ 94 cm in men and ≥ 80 cm in women
* Physical inactivity (< 2 h vigorous/active exercise training per week)

Exclusion Criteria:

* Regular use of certain prescription medications at baseline
* Severe psychiatric illness
* Pregnancy
* Pacemaker or implantable cardioverter defibrillator
* Cigarette smoking
* Previous coronary intervention
* Concomitant use of dietary supplements
* Use of omega-3 supplements at baseline
* Alcohol or drug abuse or any condition associated with poor compliance.
* Scheduled hospitalisation during the course of the study.
* Participation in a clinical trial in the last 12 weeks, or prior randomisation.
* Blood donation within the preceding 12 weeks.
* Diabetes Mellitus Type 1 or type 2
* Triglycerides > 5 mmol/l
* Previous bariatric surgery
* Malabsorption disorder

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes in lipid profile | Measured at baseline and after 8 weeks
  High-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C), total cholesterol and triglycerides (TG) will be measured in plasma/serum (mmol/L).
Changes in particle concentrations of lipoproteins of different sizes | Measured at baseline and week 8
  Particle concentration (nmol/L) of lipoprotein of different sizes will be calculated from the measured amplitude of their spectroscopically lipid methyl group NMR signals.
Changes in lipoprotein particle sizes | Measured at baseline and week 8
  Lipoprotein particle size (nm) analysis will be performed by proton nuclear magnetic resonance (NMR) spectroscopy. The size will be derived from the sum of diameter of each subclass multiplied by its relative mass percentage based on its methyl NMR signal.

SECONDARY OUTCOMES:
Changes in body composition | Measured at baseline and week 8
  Body composition will be measured by bioelectrical impedance (InBody 720).
Changes in body weight | Measured at baseline and week 8
Changes in waist and hip circumference | Measured at baseline and week 8
Changes in circulating markers of inflammation, also including adipokines and kynurenine | Measured at baseline and week 8
  Inflammatory markers and adipokines will be measured in serum/plasma, e.g tumor necrosis factor-α (TNF-α), interleukins, macrophage inflammatory protein 1-α (MIP-1-α) and granulocyte-macrophage colony stimulating factor (GM-CSF).
Changes in markers of inflammation in adipose tissue | Measured at baseline and week 8
  Inflammatory markers like TNF-α, interleukins, GM-CSF and adiponectin in will be measured in adipose tissue (pg/mg tissue).
Changes in one carbon metabolites | Measured at baseline and week 8
  Choline, betaine and related metabolites and B-vitamins involved in 1-carbon metabolism.
Changes in microbiota | Measured at baseline and week 8
  Bacterial DNA in stool samples will be subjected to high-throughput barcode multiplex sequencing of the 16s ribosomal RNA gene (rRNA).
Changes in endothelial function | Measured at baseline and week 8
  Vascular reactivity index (VRI) will be measured by monitoring fingertip temperature changes during a reactive hyperemia protocol.
Changes in carnitine and metabolites | Measured at baseline and week 8
  Trimethylamine N-oxide (TMAO), carnitine, acylcarnitines and fatty acids will be measured in serum/plasma.
Changes in gene expression in adipose tissue | Measured at baseline and week 8
  Gene expression in adipose tissue will be measured by microarray and quantitative PCR.
Changes in amino acids | Measured at baseline and week 8
  Amino acids, methylated amino acids and metabolites will be measured in serum/plasma.
Changes in gene expression i whole blood | Measured at baseline and week 8
  Gene expression in full blood will be measured by quantitative PCR.
Changes in apolipoproteins | Measured at baseline and week 8
  Apolipoproteins A1, A2, B, C2, C3 and E will be measured in serum by a multiplex kit.

CONTACTS AND LOCATIONS:
Overall Officials: Espen Rostrup, MD PhD, Principal Investigator — Haukeland University Hospital, Department of Heart Disease

REFERENCES:
- [Derived] Laupsa-Borge J, Grytten E, Bohov P, Bjorndal B, Strand E, Skorve J, Nordrehaug JE, Berge RK, Rostrup E, Mellgren G, Dankel SN, Nygard OK. Sex-specific responses in glucose-insulin homeostasis and lipoprotein-lipid components after high-dose supplementation with marine n-3 PUFAs in abdominal obesity: a randomized double-blind crossover study. Front Nutr. 2023 Jun 19;10:1020678. doi: 10.3389/fnut.2023.1020678. eCollection 2023. PMID 37404855
- [Derived] Grytten E, Laupsa-Borge J, Bohov P, Bjorndal B, Strand E, Skorve J, Nordrehaug JE, Berge RK, Rostrup E, Mellgren G, Dankel SN, Nygard OK. Changes in lipoprotein particle subclasses, standard lipids, and apolipoproteins after supplementation with n-3 or n-6 PUFAs in abdominal obesity: A randomized double-blind crossover study. Clin Nutr. 2021 May;40(5):2556-2575. doi: 10.1016/j.clnu.2021.03.040. Epub 2021 Apr 3. PMID 33933722